CLINICAL TRIAL: NCT03785249
Title: A Phase 1/2 Multiple Expansion Cohort Trial of MRTX849 in Patients With Advanced Solid Tumors With KRAS G12C Mutation KRYSTAL-1
Brief Title: Phase 1/2 Study of MRTX849 in Patients With Cancer Having a KRAS G12C Mutation KRYSTAL-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0008; CA239-0008 (Other: Bristol-Myers Squibb Protocol ID); 849-001 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2018-12-18; First posted 2018-12-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer; Metastatic Cancer; Malignant Neoplastic Disease
Keywords: KRAS; NSCLC; Colorectal Cancer; Colon Cancer; Metastatic Cancer; Pancreatic Cancer; Adagrasib; STK11 mutation; KRAS G12C
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms | interventions — adagrasib; pembrolizumab; Cetuximab; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1 Dose Exploration (Experimental): Dose escalation of MRTX849 to determine maximum tolerated dose
  Interventions: Drug: MRTX849
- Phase 1b Expansion (Experimental): Expansion cohort to ensure sufficient safety experience, pharmacokinetic information, and early evidence of clinical activity of MRTX849 to recommend Phase 2 regimens
  Interventions: Drug: MRTX849
- Phase 2 (Experimental): Separate cohorts of patients stratified by histological diagnosis, prior treatment history or co-mutation status (e.g., STK11) for evaluation of clinical activity of MRTX849
  Interventions: Drug: MRTX849
- Pilot Phase 1b Combination with Pembrolizumab (Experimental): Phase 1 evaluation of the safety, tolerability, PK and clinical activity of MRTX849 in combination with pembrolizumab in patients with NSCLC
  Interventions: Drug: MRTX849; Drug: Pembrolizumab
- Pilot Phase 1b Combination with Cetuximab (Experimental): Phase 1 evaluation of the safety, tolerability, PK and clinical activity of MRTX849 in combination with cetuximab in patients with CRC
  Interventions: Drug: MRTX849; Drug: Cetuximab
- Pilot Phase 1b Combination with Afatinib (Experimental): Phase 1 evaluation of the safety, tolerability, PK and clinical activity of MRTX849 in combination with afatinib in patients with NSCLC
  Interventions: Drug: MRTX849; Drug: Afatinib
- Phase 2 Combination with Cetuximab (Experimental): Phase 2 evaluation of the clinical activity of MRTX849 in combination with cetuximab in patients with CRC
  Interventions: Drug: MRTX849; Drug: Cetuximab
- Pilot Phase 1b Combination with Cetuximab in NSCLC (Experimental): Phase 1 evaluation of the safety, tolerability, PK and clinical activity of MRTX849 in combination with cetuximab in patients with NSCLC
  Interventions: Drug: MRTX849; Drug: Cetuximab
- Pilot Phase 1b Combination with Cetuximab in PDAC (Experimental): Phase 1 evaluation of the safety, tolerability, PK and clinical activity of MRTX849 in combination with cetuximab in patients with pancreatic adenocarcinoma (PDAC)
  Interventions: Drug: MRTX849; Drug: Cetuximab

INTERVENTIONS:
Drug: MRTX849 — MRTX849 will be administered orally once or twice daily in a continuous regimen
Drug: Pembrolizumab — Pembrolizumab is administered as an intravenous infusion once every 3 weeks
  Arms: Pilot Phase 1b Combination with Pembrolizumab
Drug: Cetuximab — Cetuximab will be administered as an intravenous infusion once per week or once every 2 weeks
  Arms: Phase 2 Combination with Cetuximab; Pilot Phase 1b Combination with Cetuximab; Pilot Phase 1b Combination with Cetuximab in NSCLC; Pilot Phase 1b Combination with Cetuximab in PDAC
Drug: Afatinib — Afatinib will be administered orally once a day in a continuous regimen
  Arms: Pilot Phase 1b Combination with Afatinib

SUMMARY:
This study will evaluate the safety, tolerability, drug levels, molecular effects, and clinical activity of MRTX849 (adagrasib) in patients with advanced solid tumors that have a KRAS G12C mutation.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, pharmacokinetics, metabolites, pharmacodynamics, and clinical activity of MRTX849 (adagrasib) in patients with advanced solid tumors with a KRAS G12C mutation. MRTX849 (adagrasib) is an orally-available small molecule inhibitor of KRAS G12C.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy with KRAS G12C mutation
* Unresectable or metastatic disease
* Standard treatment is not available or patient declines; first-line treatment for NSCLC for certain cohorts
* Adequate organ function

Exclusion Criteria:

* History of intestinal disease or major gastric surgery or inability to swallow oral medications
* Other active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety of MRTX849 in patients having advanced solid tumor malignancies with KRAS G12C mutation | 20 months
  Number of participants with treatment related adverse events
Evaluate the pharmacokinetics of MRTX849 | 20 months
  Blood plasma concentration
Evaluate clinical activity/efficacy of MRTX849 | 20 months
  Objective response rate in accordance with Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Establish maximum tolerated dose | 12 months
  Number of participants with dose limiting toxicity
Characterize safety and tolerability of MRTX849 in combination with selected therapeutic agents | 12 months
  Number of participants with dose limiting toxicity
Evaluate the pharmacokinetics of new MRTX849 oral formulations | 6 months
  Blood plasma concentration
Evaluate the pharmacokinetics of MRTX849 administered with food | 6 months
  Blood plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (222):
- United States (221):
  - Local Institution - 001-826, Birmingham, Alabama
  - Local Institution - 001-965, Anchorage, Alaska
  - Local Institution - 001-821, Phoenix, Arizona
  - Local Institution - 001-873-A, Tucson, Arizona
  - Local Institution - 001-873, Tucson, Arizona
  - Local Institution - 001-840-B, Bellflower, California
  - Local Institution - 001-834, Beverly Hills, California
  - Local Institution - 001-843, Duarte, California
  - Local Institution - 001-850-K, Dublin, California
  - Local Institution - 001-851, Fullerton, California
  - Local Institution - 001-840-C, Harbor City, California
  - Local Institution - 001-805, La Jolla, California
  - Local Institution - 001-779, Los Alamitos, California
  - Local Institution - 001-840, Los Angeles, California
  - Local Institution - 001-578, Los Angeles, California
  - Local Institution - 001-847, Newport Beach, California
  - Local Institution - 001-850-B, Oakland, California
  - Local Institution - 001-803, Orange, California
  - Local Institution - 001-850-C, Roseville, California
  - Local Institution - 001-850-J, Sacramento, California
  - Local Institution - 001-850-D, Sacramento, California
  - Local Institution - 001-845, San Diego, California
  - Local Institution - 001-840-A, San Diego, California
  - Local Institution - 001-850-H, San Francisco, California
  - Local Institution - 001-850-E, San Francisco, California
  - Local Institution - 001-850-F, San Jose, California
  - Local Institution - 001-850-A, San Leandro, California
  - Local Institution - 001-884, Santa Barbara, California
  - Local Institution - 001-850-I, Santa Clara, California
  - Local Institution - 001-884-A, Solvang, California
  - Local Institution - 001-850, Vallejo, California
  - Local Institution - 001-850-G, Walnut Creek, California
  - Local Institution - 001-872, Aurora, Colorado
  - Local Institution - 001-810, Aurora, Colorado
  - Local Institution - 001-872-H, Boulder, Colorado
  - Local Institution - 001-872-E, Colorado Springs, Colorado
  - Local Institution - 001-872-L, Colorado Springs, Colorado
  - Local Institution - 001-872-B, Denver, Colorado
  - Local Institution - 001-951 - A, Denver, Colorado
  - Local Institution - 001-951 - B, Denver, Colorado
  - Local Institution - 001-846, Grand Junction, Colorado
  - Local Institution - 001-951, Lafayette, Colorado
  - Local Institution - 001-872-A, Lakewood, Colorado
  - Local Institution - 001-872-D, Littleton, Colorado
  - Local Institution - 001-872-K, Lone Tree, Colorado
  - Local Institution - 001-872-C, Longmont, Colorado
  - Local Institution - 001-872-J, Parker, Colorado
  - Local Institution - 001-872-F, Pueblo, Colorado
  - Local Institution - 001-872-G, Pueblo, Colorado
  - Local Institution - 001-872-I, Thornton, Colorado
  - Local Institution - 001-816, New Haven, Connecticut
  - Local Institution - 001-871, Newark, Delaware
  - Local Institution - 001-929i, Altamonte Springs, Florida
  - Local Institution - 001-839, Boca Raton, Florida
  - Local Institution - 001-922A, Bonita Springs, Florida
  - Local Institution - 001-922D, Bradenton, Florida
  - Local Institution - 001-929c, Brandon, Florida
  - Local Institution - 001-922E, Cape Coral, Florida
  - Local Institution - 001-929g, Clearwater, Florida
  - Local Institution - 001-926b, Daytona Beach, Florida
  - Local Institution - 001-922, Fort Myers, Florida
  - Local Institution - 001-922B, Fort Myers, Florida
  - Local Institution - 001-922C, Fort Myers, Florida
  - Local Institution - 001-929b, Gainesville, Florida
  - Local Institution - 001-829, Jacksonville, Florida
  - Local Institution - 001-929m, Lady Lake, Florida
  - Local Institution - 001-929e, Largo, Florida
  - Local Institution - 001-929n, Lecanto, Florida
  - Local Institution - 001-870, Miami, Florida
  - Local Institution - 001-825, Miami Beach, Florida
  - Local Institution - 001-922F, Naples, Florida
  - Local Institution - 001-922G, Naples, Florida
  - Local Institution - 001-538, Ocala, Florida
  - Local Institution - 001-929p, Ocala, Florida
  - Local Institution - 001-914, Orange City, Florida
  - Local Institution - 001-929j, Orange City, Florida
  - Local Institution - 001-929l, Orlando, Florida
  - Local Institution - 001-877, Pensacola, Florida
  - Local Institution - 001-922H, Port Charlotte, Florida
  - Local Institution - 001-922I, Sarasota, Florida
  - Local Institution - 001-922J, Sarasota, Florida
  - Local Institution - 001-929h, Spring Hill, Florida
  - Local Institution - 001-929a, St. Petersburg, Florida
  - Local Institution - 001-929, St. Petersburg, Florida
  - Local Institution - 001-926d, Stuart, Florida
  - Local Institution - 001-929d, Tampa, Florida
  - Local Institution - 001-929k, Tavares, Florida
  - Local Institution - 001-929f, Trinity, Florida
  - Local Institution - 001-922K, Venice, Florida
  - Local Institution - 001-922L, Venice, Florida
  - Local Institution - 001-926c, Vero Beach, Florida
  - Local Institution - 001-926a, Wellington, Florida
  - Local Institution - 001-926, West Palm Beach, Florida
  - Local Institution - 001-929o, Winter Park, Florida
  - Local Institution - 001-967, Athens, Georgia
  - Local Institution - 001-835-C, Austell, Georgia
  - Local Institution - 001-835-E, Austell, Georgia
  - Local Institution - 001-835-D, Carrollton, Georgia
  - Local Institution - 001-835-F, Carrollton, Georgia
  - Local Institution - 001-835-A, Cartersville, Georgia
  - Local Institution - 001-835-B, Douglasville, Georgia
  - Local Institution - 001-835, Marietta, Georgia
  - Local Institution - 001-862, Chicago Ridge, Illinois
  - Local Institution - 001-883, Niles, Illinois
  - Local Institution - 001-781, South Bend, Indiana
  - Local Institution - 001-831, Iowa City, Iowa
  - Local Institution - 001-820, Westwood, Kansas
  - Local Institution - 001-844, Lexington, Kentucky
  - Local Institution - 001-920, Baton Rouge, Louisiana
  - Local Institution - 001-827, Biddeford, Maine
  - Local Institution - 001-881-B, Brandywine, Maryland
  - Local Institution - 001-881, Columbia, Maryland
  - Local Institution - 001-881-A, Silver Spring, Maryland
  - Local Institution - 001-808, Boston, Massachusetts
  - Local Institution - 001-842, Detroit, Michigan
  - Local Institution - 001-811, Detroit, Michigan
  - Local Institution - 001-842-A, Farmington Hills, Michigan
  - Local Institution - 001-838-F, Coon Rapids, Minnesota
  - Local Institution - 001-838-E, Edina, Minnesota
  - Local Institution - 001-875 - D, Edina, Minnesota
  - Local Institution - 001-838-D, Maplewood, Minnesota
  - Local Institution - 001-875 - A, Maplewood, Minnesota
  - Local Institution - 001-838-C, Minneapolis, Minnesota
  - Local Institution - 001-875, Minneapolis, Minnesota
  - Local Institution - 001-838-G, Minneapolis, Minnesota
  - Local Institution - 001-822-A, Minneapolis, Minnesota
  - Local Institution - 001-822, Minneapolis, Minnesota
  - Local Institution - 001-830, Rochester, Minnesota
  - Local Institution - 001-838, Saint Louis Park, Minnesota
  - Local Institution - 001-838-B, Saint Louis Park, Minnesota
  - Local Institution - 001-838-A, Saint Paul, Minnesota
  - Local Institution - 001-875 - B, Saint Paul, Minnesota
  - Local Institution - 001-875 - C, Woodbury, Minnesota
  - Local Institution - 001-952, Bolivar, Missouri
  - Local Institution - 001-950, Jefferson City, Missouri
  - Local Institution - 001-841, Billings, Montana
  - Local Institution - 001-544B, Omaha, Nebraska
  - Local Institution - 001-959, Omaha, Nebraska
  - Local Institution - 001-544A, Omaha, Nebraska
  - Local Institution - 001-544, Omaha, Nebraska
  - Local Institution - 001-860A, Henderson, Nevada
  - Local Institution - 001-860C, Henderson, Nevada
  - Local Institution - 001-860B, Henderson, Nevada
  - Local Institution - 001-860, Henderson, Nevada
  - Local Institution - 001-860E, Las Vegas, Nevada
  - Local Institution - 001-860D, Las Vegas, Nevada
  - Local Institution - 001-860F, Las Vegas, Nevada
  - Local Institution - 001-861, Albany, New York
  - Local Institution - 001-815, Buffalo, New York
  - Local Institution - 001-813, New York, New York
  - Local Institution - 001-806, New York, New York
  - Local Institution - 001-812, Chapel Hill, North Carolina
  - Local Institution - 001-971, Pinehurst, North Carolina
  - Local Institution - 001-966, Cincinnati, Ohio
  - Local Institution - 001-823, Cincinnati, Ohio
  - Local Institution - 001-818, Cleveland, Ohio
  - Local Institution - 001-833 - H, Columbus, Ohio
  - Local Institution - 001-833 - C, Columbus, Ohio
  - Local Institution - 001-833 - J, Columbus, Ohio
  - Local Institution - 001-833 - A, Columbus, Ohio
  - Local Institution - 001-833 - F, Columbus, Ohio
  - Local Institution - 001-833, Columbus, Ohio
  - Local Institution - 001-833 - D, Columbus, Ohio
  - Local Institution - 001-833 - I, Columbus, Ohio
  - Local Institution - 001-930, Columbus, Ohio
  - Local Institution - 001-833 - B, Columbus, Ohio
  - Local Institution - 001-833 - G, Columbus, Ohio
  - Local Institution - 001-833 - E, Gahanna, Ohio
  - Local Institution - 001-836-A, Kettering, Ohio
  - Local Institution - 001-836, Kettering, Ohio
  - Local Institution - 001-600, Lawton, Oklahoma
  - Local Institution - 001-584, Tulsa, Oklahoma
  - Local Institution - 001-586-A, Bend, Oregon
  - Local Institution - 001-586, Bend, Oregon
  - Local Institution - 001-889, Eugene, Oregon
  - Local Institution - 001-837, Allentown, Pennsylvania
  - Local Institution - 001-837-A, Bethlehem, Pennsylvania
  - Local Institution - 001-817, Hershey, Pennsylvania
  - Local Institution - 001-783, Media, Pennsylvania
  - Local Institution - 001-887, Charleston, South Carolina
  - Local Institution - 001-819, Charleston, South Carolina
  - Local Institution - 001-801-G, Gallatin, Tennessee
  - Local Institution - 001-801-A, Hendersonville, Tennessee
  - Local Institution - 001-801-D, Hermitage, Tennessee
  - Local Institution - 001-801-F, Murfreesboro, Tennessee
  - Local Institution - 001-801-B, Nashville, Tennessee
  - Local Institution - 001-801, Nashville, Tennessee
  - Local Institution - 001-801-E, Nashville, Tennessee
  - Local Institution - 001-801-C, Nashville, Tennessee
  - Local Institution - 001-888-B, Arlington, Texas
  - Local Institution - 001-888, Arlington, Texas
  - Local Institution - 001-880, Austin, Texas
  - Local Institution - 001-848a, Conroe, Texas
  - Local Institution - 001-809, Dallas, Texas
  - Local Institution - 001-886, Dallas, Texas
  - Local Institution - 001-879, Dallas, Texas
  - Local Institution - 001-785, Denison, Texas
  - Local Institution - 001-876, Fort Worth, Texas
  - Local Institution - 001-848, Houston, Texas
  - Local Institution - 001-969, Houston, Texas
  - Local Institution - 001-935A, Houston, Texas
  - Local Institution - 001-999, Irving, Texas
  - Local Institution - 001-935D, Kingwood, Texas
  - Local Institution - 001-935, Kingwood, Texas
  - Local Institution - 001-554, Midland, Texas
  - Local Institution - 001-802, San Antonio, Texas
  - Local Institution - 001-935B, Shenandoah, Texas
  - Local Institution - 001-935C, Spring, Texas
  - Local Institution - 001-874, Sugar Land, Texas
  - Local Institution - 001-935E, Tomball, Texas
  - Local Institution - 001-878, Tyler, Texas
  - Local Institution - 001-890, Waco, Texas
  - Local Institution - 001-814, Fairfax, Virginia
  - Local Institution - 001-597, Fredericksburg, Virginia
  - Local Institution - 001-882, Newport News, Virginia
  - Local Institution - 001-882-A, Norfolk, Virginia
  - Local Institution - 001-890-A, Norfolk, Virginia
  - Local Institution - 001-968, Richmond, Virginia
  - Local Institution - 001-824, Seattle, Washington
  - Local Institution - 001-885, Vancouver, Washington
  - Local Institution - 001-804, Madison, Wisconsin
- Local Institution - 001-900, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Negrao MV, Spira AI, Heist RS, Janne PA, Pacheco JM, Weiss J, Gadgeel SM, Velastegui K, Yang W, Der-Torossian H, Christensen JG, Sabari JK. Intracranial Efficacy of Adagrasib in Patients From the KRYSTAL-1 Trial With KRASG12C-Mutated Non-Small-Cell Lung Cancer Who Have Untreated CNS Metastases. J Clin Oncol. 2023 Oct 1;41(28):4472-4477. doi: 10.1200/JCO.23.00046. Epub 2023 Jun 16. PMID 37327468
- [Derived] Bekaii-Saab TS, Yaeger R, Spira AI, Pelster MS, Sabari JK, Hafez N, Barve M, Velastegui K, Yan X, Shetty A, Der-Torossian H, Pant S. Adagrasib in Advanced Solid Tumors Harboring a KRASG12C Mutation. J Clin Oncol. 2023 Sep 1;41(25):4097-4106. doi: 10.1200/JCO.23.00434. Epub 2023 Apr 26. PMID 37099736
- [Derived] Yaeger R, Weiss J, Pelster MS, Spira AI, Barve M, Ou SI, Leal TA, Bekaii-Saab TS, Paweletz CP, Heavey GA, Christensen JG, Velastegui K, Kheoh T, Der-Torossian H, Klempner SJ. Adagrasib with or without Cetuximab in Colorectal Cancer with Mutated KRAS G12C. N Engl J Med. 2023 Jan 5;388(1):44-54. doi: 10.1056/NEJMoa2212419. Epub 2022 Dec 21. PMID 36546659
- [Derived] Janne PA, Riely GJ, Gadgeel SM, Heist RS, Ou SI, Pacheco JM, Johnson ML, Sabari JK, Leventakos K, Yau E, Bazhenova L, Negrao MV, Pennell NA, Zhang J, Anderes K, Der-Torossian H, Kheoh T, Velastegui K, Yan X, Christensen JG, Chao RC, Spira AI. Adagrasib in Non-Small-Cell Lung Cancer Harboring a KRASG12C Mutation. N Engl J Med. 2022 Jul 14;387(2):120-131. doi: 10.1056/NEJMoa2204619. Epub 2022 Jun 3. PMID 35658005
- [Derived] Sabari JK, Velcheti V, Shimizu K, Strickland MR, Heist RS, Singh M, Nayyar N, Giobbie-Hurder A, Digumarthy SR, Gainor JF, Rajan AP, Nieblas-Bedolla E, Burns AC, Hallin J, Olson P, Christensen JG, Kurz SC, Brastianos PK, Wakimoto H. Activity of Adagrasib (MRTX849) in Brain Metastases: Preclinical Models and Clinical Data from Patients with KRASG12C-Mutant Non-Small Cell Lung Cancer. Clin Cancer Res. 2022 Aug 2;28(15):3318-3328. doi: 10.1158/1078-0432.CCR-22-0383. PMID 35404402
- [Derived] Ou SI, Janne PA, Leal TA, Rybkin II, Sabari JK, Barve MA, Bazhenova L, Johnson ML, Velastegui KL, Cilliers C, Christensen JG, Yan X, Chao RC, Papadopoulos KP. First-in-Human Phase I/IB Dose-Finding Study of Adagrasib (MRTX849) in Patients With Advanced KRASG12C Solid Tumors (KRYSTAL-1). J Clin Oncol. 2022 Aug 10;40(23):2530-2538. doi: 10.1200/JCO.21.02752. Epub 2022 Feb 15. PMID 35167329
- [Derived] Awad MM, Liu S, Rybkin II, Arbour KC, Dilly J, Zhu VW, Johnson ML, Heist RS, Patil T, Riely GJ, Jacobson JO, Yang X, Persky NS, Root DE, Lowder KE, Feng H, Zhang SS, Haigis KM, Hung YP, Sholl LM, Wolpin BM, Wiese J, Christiansen J, Lee J, Schrock AB, Lim LP, Garg K, Li M, Engstrom LD, Waters L, Lawson JD, Olson P, Lito P, Ou SI, Christensen JG, Janne PA, Aguirre AJ. Acquired Resistance to KRASG12C Inhibition in Cancer. N Engl J Med. 2021 Jun 24;384(25):2382-2393. doi: 10.1056/NEJMoa2105281. PMID 34161704
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03785249.html